CLINICAL TRIAL: NCT03789630
Title: Observation of In-home Continuous Monitoring of Human Physiology and Self-reported Pain Score Among Knee Replacement, Anterior Cruciate Ligament (ACL), Knee Arthroscopy & Foot & Ankle Related Surgery Patients
Brief Title: Continuous Monitoring of Physiology and Self-reported Pain Score Amongst Post-surgical Knee Patients
Acronym: ObservePAIN
Status: Completed | Type: Observational
Sponsor: Biofourmis Singapore Pte Ltd. (Industry)
Collaborators: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CT002
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Knee Arthroplasty
Keywords: Knee Replacement; Wearable; Pain Score Quantification
MeSH Terms: interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Monitoring arm: Monitoring subjects undergoing total knee replacement surgery using the wearable biosensor to continuously monitor physiology biomarkers.
  Interventions: Device: Continuous physiology monitoring in ambulatory setting pre and post surgery

INTERVENTIONS:
Device: Continuous physiology monitoring in ambulatory setting pre and post surgery — This study will recruit 55 patients aged 21 to 80 years who will be undergoing total knee replacement surgery. All study participants undergoing total knee replacement surgery will be monitored using the wearable biosensor to continuously monitor physiology biomarkers. Participants will be followed for an estimated total of 39 days, beginning four days before surgery, the entire period during in-patient recovery (four to five days), and 30-days post-discharge at-home.

SUMMARY:
The aim of this observational study is to assess whether patient reported pain levels correlate with a Pain Index derived from deviations in multivariate physiology biomarkers captured in real-world setting. This study will be conducted using a clinical-grade wearable sensor to continuously monitor patient's physiology (pain related biomarkers) and allow subject participant to actively report their pain score, symptoms and quality of life using a mobile-based application.

DETAILED DESCRIPTION:
The designated clinical-grade wearable sensor used in this study is the Biovotion Everion MD (See Annex for product description), a Bluetooth-compatible device that will automatically sync with the mobile application used in this study.

This study will recruit 55 patients aged 21 to 80 years who will be undergoing knee replacement, Anterior Cruciate Ligament(ACL), Knee Arthroscopy and Foot & Ankle related surgery. All study participants will be followed for an estimated total of 30 days(+6/-2 days, if visit schedule is fall on weekend), beginning four days before surgery, the entire period as an in-patient (four to five days), and 20-days post-discharge.

The changes in multivariate physiological biomarkers will be used to generate a Pain Index, and the Pain Index will be assessed against patient reported Numerical Rating Scale (NRS) pain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 21 to 80 years
* Patients undergoing knee replacement surgery ( Total Knee Replacement (TKR), Unicompartmental Knee arthroplasty (UKA), Bilateral knee replacemenent, Patello-Femoral-Joint (PFJ) Knee replacement), Anterior Cruciate Ligament(ACL), Knee Arthroscopy and Foot & Ankle related surgery such as bunions, hammer toes, metatarsal, ankle fusion, triple fusion, ankle replacement, achilles tendon & tibialis posterior disorder
* Ability to provide informed consent
* Able to commit to using the app and inputting data as needed during the study duration
* Has access to an iPhone (minimum requirement iPhone 5S)

Exclusion Criteria:

* Previous myocardial infarction (MI)
* Known coronary artery disease - prior coronary revascularization
* Previous stroke. Stroke is defined as new focal neurological deficit perspective more than 24 hours.
* More than ongoing use of 2 or more anti-hypertensive agents.
* Expected life expectancy less than 1 year.
* Asthma or chronic lung disease requiring long-term medications or oxygen
* Mental illness that in the clinical judgment of the investigator will affect participation in the study e.g. dementia
* Inability to comply with the study protocol
* Any other acute or chronic medical or physical condition deemed by the investigator to affect study outcomes

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 55 study participants, aged between 21 to 80 years, regardless of gender, who is undergoing total knee replacement surgery will be enrolled for the study upon receiving informed consent.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Pain Correlation (using binary pain classification) | 30 days
  Agreement between patient-reported NRS pain (classified into None-Mild and Moderate-Severe) and Pain Index, measured using Kappa statistic.

SECONDARY OUTCOMES:
Pain Correlation in Opioid Medication Subgroup | 30 days
  Agreement between patient-reported NRS pain and Pain Index in patients using opioid medication for post-surgical pain relief, measured using Kappa statistic.
Pain Correlation (3 pain categories) | 30 days
  Agreement between patient-reported NRS pain (classified into None-Mild, Moderate and Severe) and Pain Index, measured using Kappa statistic.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital (SGH), Singapore, Singapore